CLINICAL TRIAL: NCT06929988
Title: A Clinical Safety, In-use Tolerability and Efficacy Study of the Test Product in Heathy Adult Human Subjects With Dry or Sensitive Skin
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Test Product in Healthy Adult Human Subjects With Dry or Sensitive Skin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SAVA Healthcare Limited (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB250005-SG
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Dry Skin; Sensitive Skin

STUDY DESIGN:
Intervention Model Description: Test Product A: Creanz Lotion Mode of Usage: Apply sufficient quantity of Creanz Nourishing Body lotion to face and body for smooth and moisturised skin.
  Frequency: Twice a Day Route of Administration: Topical
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Creanz Lotion (Experimental): Mode of Usage: Apply sufficient quantity of Creanz Nourishing Body lotion to face and body for smooth and moisturised skin.
  Frequency: Twice a Day Route of Administration: Topical
  Interventions: Other: Creanz Lotion

INTERVENTIONS:
Other: Creanz Lotion — Mode of Usage: Apply sufficient quantity of Creanz Nourishing Body lotion to face and body for smooth and moisturised skin.
  Frequency: Twice a Day Route of Administration: Topical

SUMMARY:
This exploratory, prospective, open-label, single-centre, safety, efficacy and in-use tolerability study of the test product in healthy adult human subjects with dry or sensitive skin.

DETAILED DESCRIPTION:
A total of up to 32 healthy male and non-pregnant | non-lactating female with dry or sensitive skin and an age of 18-55 years will be enrolled to complete the 30 subjects of the study.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called telephonically by the recruiting department prior to the enrollment visit. Subjects will be told during screening (prior to enrolment) not to wear any facial make-up on the study visit day. The adult female subjects will be instructed to visit the facility as per the below visits.

Visit 01 (Day 01): Screening, Enrolment, Baseline Evaluation, On Site Product Usage, Post Usage Evaluation Visit 02 (Day 02): Evaluations, Product usage period Visit 03 (Day 15 +2 Days): Evaluations, End of the Study

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 55 years (both inclusive) at the time of consent.
* Sex: Healthy male and non-pregnant/non-lactating females.
* Females of childbearing potential must have a self-reported negative pregnancy test.
* Subject are generally in good health.
* Subject with dry or sensitive skin at a time of screening. (Dermatological Assessment)
* Subjects assessment site must be free of cuts, tattoos, scratches, abrasions, scars, uneven skin tone, sunburn, excessive tan, excessive hair or open wounds.
* Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
* If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
* Subjects are willing to give written informed consent and are willing to come for regular follow up.
* Subjects who commit not to use medicated skincare products other than the test product for the entire duration of the study.
* Subject who have not participated in a similar investigation in the past three months.
* Willing to use test product throughout the study period.

Exclusion Criteria:

* History of any dermatological condition of the skin diseases.
* Subject with present condition of allergic response to any cosmetic product.
* Subject having allergic response to the ink.
* Presence of any broken, chapped, cut, irritated, or scraped skin at the application site.
* Subjects under chronic medication (e.g. aspirin-based products, anti-inflammatories, anti-histamines, corticotherapy etc.) that might influence the outcome of the study.
* Subject having acne of severe incidence (presence of nodules, cysts or numerous pustules) which requires pharmaceutical or cosmeceuticals, herbal treatment.
* Subjects who have applied topical treatment for at least 4 weeks and any systemic treatment for at least 3 months, before they participated in the study.
* History of alcohol or drug addiction.
* Subjects using other marketed products during the study period.
* Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
* Pregnant or breastfeeding or planning to become pregnant during the study period.
* History of chronic illness which may influence the cutaneous state.
* Subjects participating in other similar cosmetics, devices or therapeutic trials or skincare products within the last four weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in skin hydration | baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Instrumental Assessment: Corneometer CM 825
Change in skin elasticity | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Instrumental Assessment: Cutometer Dual MPA 580
Change in Dry skin area and severity index | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological assessment: 0 = Absent; 4 = Severe
Change in Overall Dry skin Score | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological assessment: 0 = Absent; 4 = Dominated by large scales
Change in skin barrier function | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Instrumental Assessment: TEWAMeter TM Hex
Change in skin roughness | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Instrumental Assessment: VISIOSCAN VC 20 Plus
Change in skin scaliness | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Instrumental Assessment: VISIOSCAN VC 20 Plus
Change in skin smoothness | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Instrumental Assessment: VISIOSCAN VC 20 Plus
Change in skin wrinkles | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Instrumental Assessment: VISIOSCAN VC 20 Plus

SECONDARY OUTCOMES:
Change in itchiness score | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological Assessment: VAS score 0= no itch,10 = severe itch
change in visual assessment of skin dryness, | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological Assessment: 0= absent,4 = Extreme
Change in visual assessment of skin smoothness, | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological Assessment: 0= absent,4 = severe
Change in visual assessment of skin roughness, | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological Assessment: 0= absent,4 = extreme
Change in visual assessment of skin scaliness, | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological Assessment: 0= absent,4 = extreme
Change in visual assessment of skin redness, | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological Assessment: 0= absent,4 = extreme
Change in visual assessment of skin itchiness | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Dermatological Assessment: 0= None,4 = severe
Change in product perception Questionnaire | Baseline before usage of the test product on Day 01 and after usage of the test product at T20 mins on Day 01, Day 02, and Day 15 (+2 Days)
  Scoring scale: 9-point hedonic scale

CONTACTS AND LOCATIONS:
Overall Officials: Nayan Patel, MBBS, Principal Investigator — NovoBliss Research Private Limited
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No